CLINICAL TRIAL: NCT06321445
Title: The Success of ChatGPT in Providing American Society of Anesthesiologist (ASA) Scores
Acronym: ASA
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ChatGptASAscore
Record Dates: First submitted 2024-03-11; First posted 2024-03-20 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Artificial Intelligence; Preoperative Evaluation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experts: ASA scores provided by anesthesiologists
  Interventions: Other: providing ASA score
- ChatGpt: ASA scores provided by ChatGpt
  Interventions: Other: providing ASA score

INTERVENTIONS:
Other: providing ASA score — ASA scoring, or the American Society of Anesthesiologists (ASA) Physical Status Classification System, is a framework used by anesthesiologists to assess the preoperative physical fitness of a patient before surgery. It categorizes patients into six classes based on their overall health status, ranging from ASA I (a healthy patient) to ASA VI (a declared brain-dead patient whose organs are being removed for donor purposes). The ASA score helps in predicting perioperative risks and assists healthcare professionals in making informed decisions about anesthesia management and the need for special precautions during and after surgery.

SUMMARY:
Patients applied to the anesthesia clinics of Health Science University Istanbul Kanuni Sultan Suleyman Training and Research Hospital and Basaksehir Cam and Sakura City Hospital were included in the study. Evaluation forms which will be filled in every preoperative examinations will be saved in the hospitals systems. Patients datas without indentification informations will be asked to ChatGpt to give anesthesiological risc scores. This scores will be compared with the scores already given by anesthesiologists.

DETAILED DESCRIPTION:
Patients of all ages and sexes with ASA scores ranging from I to IV who applied to the anesthesia clinics of Health Science University Istanbul Kanuni Sultan Suleyman Training and Research Hospital and Basaksehir Cam and Sakura City Hospital were included in the study. Patients with ASA scores of V and VI were not included in the study as their statistical distribution would be disrupted.

Data Collection Data were collected daily from preoperative examination evaluation forms in this study, which included Patient's Age Patient's Gender Patient's Weight Patient's Height Additional Illnesses Medications Used Abnormal Laboratory Findings Abnormal Imaging Findings Operation to be Performed Consultation Notes Given ASA Score ChatGPT's ASA Score. At Health Science University Istanbul Kanuni Sultan Suleyman Training and Research Hospita, the patient will be under the care of Specialist Doctor Engin İhsan Turan, and at Basaksehir Cam and Sakura City Hospital, under the care of Specialist Doctor Abdurrahman Engin Baydemir.

The natural language processing module ChatGPT 4, developed by OpenAI, was consulted for providing ASA scores based on the collected data. In addition to the collected data, ASA scores given by anesthesia experts were also entered into the system.

The investigators chose ChatGPT-4 among artificial intelligence models for our study due to its extensive use in the literature.

Primary Objective: To evaluate the success of ChatGPT-4 in predicting postoperative intensive care needs and mortality in adult patients with ASA scores of III and IV. Secondary Objectives: To examine the effectiveness of ChatGPT-4's recommendations on anesthesia methods and additional suggestions in the clinical decision-making process.

Benefits: Understanding the contributions of artificial intelligence-based systems to clinical decision-making processes.

Risks: The potential for ChatGPT-4's recommendations to be misleading, but the risk will be mitigated by doctors being the final decision-makers.

Use of ChatGPT 4 After the data mentioned above regarding the patients were transmitted to ChatGPT 4, ChatGPT 4 was asked to predict the ASA scores of the patients. To do so the investigators will create a special GPT which can provide ASA scores according to the newest guidelines. This GPT will assign patients an ASA score based on abnormal data while recognizing that the patients' other results and physical examination findings are normal.

ELIGIBILITY:
Inclusion Criteria:

* Patient who admitted to anesthesia clinics for both hospital
* Patient with ASA scores between I-IV

Exclusion Criteria:

* ASA scores higher than IV
* Emergency cases patients have symptoms like upper and lower airway infections.
* patients haven't got enough informations to provide ASA scores.
* Patients with symptoms of an active upper or lower respiratory tract infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who admitted to anesthesia clinics of Health Science University Istanbul Kanuni Sultan Suleyman Training and Research Hospital and Basaksehir Cam and Sakura City Hospital.
Sampling Method: Probability Sample
Enrollment: 2851 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The Success of ChatGPT in Providing American Society of Anesthesiologist (ASA) Scores | 2 weeks
  Comparison of ASA scores provided from ChatGpt and provided from anesthesiologists.
  ASA 1: A normal healthy patient. ASA 2: A patient with mild systemic disease. ASA 3: A patient with severe systemic disease that is not incapacitating. ASA 4: A patient with severe systemic disease that is a constant threat to life.
  ASA 5: A moribund patient who is not expected to survive without the operation. ASA 6: A declared brain-dead patient whose organs are being removed for donor purposes.
  Additional classifications include:
  E: This designation can be added to any of the above classifications (ASA 1E to ASA 6E) to indicate that the surgery is an emergency, which increases the risk of the procedure.

SECONDARY OUTCOMES:
The Success of ChatGPT in clinical decisions | 2 weeks
  Comparison of ASA scores provided from ChatGpt and provided from anesthesiologists.
  ASA 1: A normal healthy patient. ASA 2: A patient with mild systemic disease. ASA 3: A patient with severe systemic disease that is not incapacitating. ASA 4: A patient with severe systemic disease that is a constant threat to life.
  ASA 5: A moribund patient who is not expected to survive without the operation. ASA 6: A declared brain-dead patient whose organs are being removed for donor purposes.
  Additional classifications include:
  E: This designation can be added to any of the above classifications (ASA 1E to ASA 6E) to indicate that the surgery is an emergency, which increases the risk of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yeo YH, Samaan JS, Ng WH, Ting PS, Trivedi H, Vipani A, Ayoub W, Yang JD, Liran O, Spiegel B, Kuo A. Assessing the performance of ChatGPT in answering questions regarding cirrhosis and hepatocellular carcinoma. Clin Mol Hepatol. 2023 Jul;29(3):721-732. doi: 10.3350/cmh.2023.0089. Epub 2023 Mar 22. PMID 36946005
- [Result] Wongtangman K, Aasman B, Garg S, Witt AS, Harandi AA, Azimaraghi O, Mirhaji P, Soby S, Anand P, Himes CP, Smith RV, Santer P, Freda J, Eikermann M, Ramaswamy P. Development and validation of a machine learning ASA-score to identify candidates for comprehensive preoperative screening and risk stratification. J Clin Anesth. 2023 Aug;87:111103. doi: 10.1016/j.jclinane.2023.111103. Epub 2023 Mar 8. PMID 36898279
- [Derived] Turan EI, Baydemir AE, Ozcan FG, Sahin AS. Evaluating the accuracy of ChatGPT-4 in predicting ASA scores: A prospective multicentric study ChatGPT-4 in ASA score prediction. J Clin Anesth. 2024 Sep;96:111475. doi: 10.1016/j.jclinane.2024.111475. Epub 2024 Apr 23. PMID 38657530